CLINICAL TRIAL: NCT05687201
Title: Effect of Apolipoprotein E4 on Perihematomal Edema and Short-term Prognosis in Patients With Intracerebral Hemorrhage
Brief Title: Effect of Apolipoprotein E on the Prognosis of Patients With Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Lei Huang, Principal Investigator, The Affiliated Hospital Of Guizhou Medical University
Other Study IDs: HL970570
Record Dates: First submitted 2022-12-21; First posted 2023-01-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Apolipoprotein E gene; Perihematomal edema; Outcome
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APOE-E4 (ε2/ε4,ε3/ε4,ε4/ε4) group: All the patients in this study received the same medications based on the guidelines for the management of hypertensive intracerebral hemorrhage.In addition, all patients received more comprehensive measures to prevent deep vein thrombosis (DVT), control blood pressure and glucose, nutritional support, and prevent other complications.
  Interventions: Diagnostic Test: Non-enhanced CT scan、Nuclear Magnetic Resonance (MRI)
- APOEε3(ε3/ε3) group: All the patients in this study received the same medications based on the guidelines for the management of hypertensive intracerebral hemorrhage.In addition, all patients received more comprehensive measures to prevent deep vein thrombosis (DVT), control blood pressure and glucose, nutritional support, and prevent other complications.
  Interventions: Diagnostic Test: Non-enhanced CT scan、Nuclear Magnetic Resonance (MRI)

INTERVENTIONS:
Diagnostic Test: Non-enhanced CT scan、Nuclear Magnetic Resonance (MRI) — Non-surgical patients were followed up by CT on days 1 and 5-7 after ICH, and by CT or MRI on day 5-7. Surgical patients were followed up by CT before surgery and then transferred to the operating room. The first postoperative follow-up CT scan was performed on the second day after surgery, and the second postoperative CT scan was performed on the third day after surgery. Some patients need a third or even a fourth CT follow-up after surgery. The CT scan can be repeated at any time if the patient has neurologic deterioration.

SUMMARY:
The purpose of this observational study was to compare perihematomal edema and short-term prognosis in patients with intracerebral hemorrhage carrying the APOE-ε3 and APOE-ε4 genes. The main questions it aims to answer are:

* Exploring whether patients carrying the ApoE-ε4 gene have more perifocal perihematomal edema after intracerebral hemorrhage than patients with the ApoE-ε3 gene.
* ApoEε4 gene has worse short-term prognosis than ApoEε3 gene in intracerebral hemorrhage patients.

All the patients in this study received the same medications based on the guidelines for the management of hypertensive intracerebral hemorrhage.Some ICH patients were evaluated for Stereotactic minimally invasive surgery (sMIS) treatment by two experienced neurosurgeons.

ELIGIBILITY:
Inclusion Criteria:

* Relevant diagnosis of supratentorial ICH was confirmed through unenhanced CT scanning.
* Patients were distinguished based on venous blood collection, with the presence of the ApoE-ε4 (ε2/ε4, ε3/ε4, ε4/ε4) gene (ApoE-ε4 genotype) and patients harboring the ApoE-ε3 (ε3/ε3) gene (non-ApoE-ε4 genotype).

Exclusion Criteria:

* Patients with infratentorial ICH.
* Patients with ApoE-ε2 (ε2/ε2) based on venous blood collections.
* Younger than 18 years of age.
* ICH caused by trauma, anticoagulation therapy, or antiplatelet therapy.
* Patients admitted to the hospital with diseases that might impact inflammatory responses, such as infective meningitis and systemic infections.
* Patients with previous residual neurological deficits following a stroke.
* Patients with combined tumours, severe liver and kidney dysfunction, cardiac insufficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective cohort study on spontaneous ICH was conducted at the Affiliated Hospital of Guizhou Medical University from January 2020 to December 2023. The patients were diagnosed with ICH by CT scan and has APOE gene test results. Screening was performed according to the following inclusion criteria, and patients meeting the above criteria were divided into ApoE-ε3 and ApoE-ε4 groups according to APOE test results.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
One month after ICH | A maximum of 1 month was assessed from the date of randomization to the date of the first record of progression or death from any cause, whichever came first.
  Telephone follow-up by experienced neurologist.Defining a modified Rankin Scale (mRS) score of 0-3 at discharge was considered to be a good prognosis. If the mRS score was >3, the prognosis was considered poor.
Volume of perihematoma edema | Within 24 hours of ICH
  Calculation of perihematoma edema volume after ICH by non-enhanced CT scan.
Changes in the volume of perihematoma edema | Days 5-7 after ICH
  Calculation of perihematoma edema volume after ICH by non-enhanced CT scan.

SECONDARY OUTCOMES:
Venous blood indicators | Within 24 hours of the onset of ICH
  Indicators of venous blood leukocytes, neutrophils and blood lymphocytes (10^9/L) were analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Computed Tomography, Guiyang, Guizhou, China

REFERENCES:
- [Derived] Huang L, Wu Q, Ye F, Che W, Zhao X, Yang C, Ren S, Wu G, Wang L. Apolipoprotein E-epsilon4 allele is associated with perihematomal brain edema and poor outcomes in patients with intracerebral hemorrhage. Sci Rep. 2025 Feb 16;15(1):5682. doi: 10.1038/s41598-025-89868-3. PMID 39956815